CLINICAL TRIAL: NCT03396900
Title: Periodontally Accelerated Osteogenic Orthodontics Combined With Recombinant Human Bone Morphogenetic Protein-2: An Outcome Assessment
Brief Title: Periodontally Accelerated Osteogenic Orthodontics With BMP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/2/2015
Record Dates: First submitted 2017-12-27; First posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion | interventions — recombinant human bone morphogenetic protein-2

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled clinical trial where systemically healthy individuals undergoing orthodontic therapy and willing to participate in the study were referred from the Department of Orthodontics and were followed up over a 6 month period after treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The orthodontist (HA) who performed the relevant treatment after PAOO was different from the orthodontist (MRR) randomizing the subjects into C or C+BMP groups and hence was blinded to the treatment received by the patient. One periodontist performed the PAOO surgeries (KM) and another periodontist (RVC) blinded to the therapy received by the subjects recorded the clinical and radiographic data pertinent to the study. The blind was not broken until the end of study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RhBMP-2 Protein, Recombinant (Active Comparator): 15 subjects treated with corticotomy with rhBMP-2 (C+BMP)
  Interventions: Drug: RhBMP-2 Protein, Recombinant
- Conventional Corticotomy (Experimental): 15 subjects treated with conventional corticotomy (C) as in the PAOO protocol
  Interventions: Other: Conventional Corticotomy

INTERVENTIONS:
Drug: RhBMP-2 Protein, Recombinant — Bone morphogenetic proteins (BMPs) are a category of proteins that are involved in bone formation and repair. Among these, BMP-2 is one of the most potent members of the BMP family and has been used for correcting intrabony, supraalveolar, furcation, and fenestration defects due to its osteoinductive property. BMP's are also essential for differentiation of osteoclasts, but their role in this process remains unclear. Treatment of osteoclasts with exogenous BMP-2 directly enhances RANKL-stimulated differentiation of osteoclast precursors in vitro and stimulates survival and resorptive activity of mature osteoclasts that accelerates the tooth movement.
  Other Names: Osteogenic protein
  Arms: RhBMP-2 Protein, Recombinant
Other: Conventional Corticotomy — A conventional PAOO Surgical procedure will be performed for individuals in this arm
  Other Names: PAOO Surgery
  Arms: Conventional Corticotomy

SUMMARY:
rhBMP-2 has the potential to function as a regenerative material in periodontally accelerated osteogenic orthodontics (PAOO). This study aimed to assess the effects of PAOO with BMP-2 on outcomes such as treatment period, bone density, healing and pain.

DETAILED DESCRIPTION:
Subjects were randomly assigned into each of the following experimental groups; C+BMP: corticotomy with 0.5 μg/mL rhBMP-2 and C: corticotomy only. Clinical parameters included recording the duration of treatment period, visual analogue scale (VAS) scores and early healing index (EHI) scores. The evaluation of bone density was performed at baseline, 3 months and 6 months by using RVG.

ELIGIBILITY:
Inclusion Criteria:

* 30 subjects with moderate crowding of lower incisors based upon Little's index and willing to undergo undergoing orthodontic treatment with extraction therapy of lower 1st premolars and PAOO were included in the study.

Exclusion Criteria:

* Smokers and subjects with severe crowding of anterior teeth, periodontitis and systemic diseases were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Orthodontic treatment duration | Up to 6 months
  Periodic recall of patients for every two weeks was done to assess the amount of crowding relieved by using digital Vernier calipers and photographs. The time taken to unravel the crowding in the pretreatment and post treatment study models and photographs was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar R Rachala, MDS, Study Chair — SVS Institute of Dental Sciences
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Published data will be shared